CLINICAL TRIAL: NCT01442467
Title: Correlation Between Echocardiographic Indices of Diastolic Function (E/E') and Left Ventricular End Diastolic Pressure (LVEDP) in Patients With Mitral Annular Calcification
Brief Title: Study of Echocardiogram Accuracy in Patients With Mitral Valve Calcification
Status: Terminated | Type: Observational
Why Stopped: Subject accrual too difficult
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: 11-16085
Record Dates: First submitted 2011-08-08; First posted 2011-09-28 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-03

CONDITIONS: Mitral Annulus Calcification
Keywords: mitral annular calcification; MAC; left atrial pressure; LAP; left ventricular end diastolic pressure; LVEDP; Echocardiogram

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mild to Severe MAC
- No to mild MAC

SUMMARY:
This study aims to evaluate the accuracy of the echocardiographic data obtained from patients with calcifications in the mitral valve who are undergoing a cardiac (heart) catheterization.

Echocardiography is a non-invasive (does not break the skin) procedure used to see an image of the heart. It uses harmless sound waves to create an image of the heart on a computer screen. These images will show the valves of the heart, how well the heart is pumping blood, the blood flow across these valves and how large the heart is. A silver paddle-shaped device is moved easily over the skin to capture these images.

Calcification (hardening) of the heart valves and heart rings (fibrous tissue surrounding the valves) is a common finding and it increases with age. The presence of calcification changes the blood flow through the heart valves. This makes any echocardiographic data (information) obtained from patients with calcifications difficult to interpret.

DETAILED DESCRIPTION:
Patients with significant mitral annular calcification (MAC) have largely been excluded from studies validating non invasive (echocardiographic) measurements of left ventricular filling and diastolic function. The investigators hypothesize that echocardiographic estimates of diastolic function, left atrial pressure (LAP) and left ventricular end diastolic pressure (LVEDP) are likely to be fallacious in patients with moderate to severe mitral annular calcification due to the structural alterations and technical difficulties involved.

ELIGIBILITY:
Inclusion Criteria:

* >= 19 years of age
* undergoing planned cardiac catheterization

Exclusion Criteria:

* < 19 years of age
* acute coronary syndrome
* decompensated heart failure
* not in sinus rhythm
* > mild MR
* hypertensive urgency/emergency
* severe aortic stenosis
* poor echo windows for Doppler imaging

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elective/planned cardiac catheterization
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Agreement between invasive and non-invasive measures of LVEDP | participants will be followed for the duration of hospital stay, an expected average of 2 days
  evaluate the agreement between the E/E' ratio by echocardiography and the left ventricular end-diastolic pressure by cardiac catheterization in patients with moderate to severe mitral annular calcification

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton Unviversity Medical Center, Omaha, Nebraska, United States